CLINICAL TRIAL: NCT06407349
Title: Effect of Communication Board on Functional Communication of Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01777 Imtasha Rana
Record Dates: First submitted 2024-04-29; First posted 2024-05-09 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Cerebral Palsy (CP)
MeSH Terms: conditions — Cerebral Palsy | interventions — Communication Devices for People with Disabilities

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Communication Board (Experimental): customized individualized AAC communication Board with a step command Intervention description: 3 sessions per week, of 30 minutes total of 24 sessions. Both genders will be included.
  Children's ages range from 8 to 12 years.
  Interventions: Other: Communication Board
- Traditional Therapy (Other): Traditional therapy with one-step command Intervention description: 3 sessions per week, of 30 minutes total of 24 sessions. Both genders will be included.
  Children's ages range from 8 to 12 years.
  Interventions: Other: Traditional Therapy

INTERVENTIONS:
Other: Communication Board — communication board based on a functional communication picture of basic needs of categories ( food, clothes, object, and actions)
  Arms: Communication Board
Other: Traditional Therapy — Traditional Therapy
  Arms: Traditional Therapy

SUMMARY:
My aim of the research is to compare the effect of traditional therapy with the AAC device and identify if the AAC device is more effective for CP children than traditional therapy.

ELIGIBILITY:
Inclusion Criteria:

* Children of both genders with Cerebral Palsy age group 8 years-12 years
* Children with Cerebral Palsy having mild to moderate cognitive impairment and communication impairment
* Children with comorbid conditions (epilepsy, microcephalia)
* Children with physical abilities of functional Pointing, One Step Command
* Following, Vocalization, and Imitation.

Exclusion Criteria:

* Children with comorbid conditions (visual impairment, hearing impairment

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Functional Communication | 8th week
  Baseline measurement of all the individuals who are enrolled in the study will be taken by using the following assessment tools.
  Functional communication checklist; provide the score with reference to five domains- method of communication, communication interaction, communication function, expressive language skills, and receptive language skills Communication effective index will also be used which consists of sixteen items.
  Information Carrying words will be used based on age. After baseline measurements communication board intervention will be given to the individuals with cerebral palsy belonging to the experimental group while traditional therapy will be given to the control group. After providing the mentioned treatment to both groups for twenty four sessions, the post-assessment will be taken.

CONTACTS AND LOCATIONS:
Overall Officials: Maimoona Ismail, Principal Investigator — Riphah International University
Locations (1):
- Special Education Academy, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No